CLINICAL TRIAL: NCT01629030
Title: Risk Factors of Sternal Wound Infection After Coronary Artery Bypass Graft
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sangmin M. Lee, Professor, Samsung Medical Center
Other Study IDs: 2012-05-067-001
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Coronary Artery Bypass Graft; Median Sternotomy
Keywords: sternal wound infection; coronary artery bypass graft; risk factor

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coronary Artery Bypass Graft Group: Those underwent coronary artery bypass graft surgery with median sternotomy in Samsung Medical Center during the period of January 2008 and December 2011.

SUMMARY:
The investigators are trying to evaluate the performance of neutrophil and lymphocyte counts as a risk factor of deep sternal wound infection after coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
Deep sternal wound infection after coronary artery bypass graft is a very dangerous complication as it prolongs hospital stay, increase morbidity and mortality, and increase cost of care.

As a risk factor of surgical site infection, risk index reported by NNIS (national nosocomial infection surveillance), Euroscore, or Society of thoracic surgeon risk score are currently used. However, as various performances are reported regarding these index or scoring systems, and many factors are needed for these index or scoring system, there is a need to develop a more simple risk factor with better performance. We focused on the differential blood cell count, as the neutrophil and lymphocyte count are related to the degree of surgical invasion, and inflammatory response. Previous studies reported that the neutrophilia or lymphopenia is related to postoperative infection. Therefore, we are trying to evaluate the performance of preoperative or postoperative the blood cell differential count as a risk factor for sternal wound infection after coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Those underwent coronary artery bypass graft surgery with median sternotomy in Samsung Medical Center during the period of January 2008 and December 2011.

Exclusion Criteria:

* Those underwent coronary artery bypass graft surgery with mini-thoracotomy
* Those with insufficient study data recognized by electronic medical record

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those underwent coronary artery bypass graft surgery with median sternotomy in Samsung Medical Center during the period of January 2008 and December 2011.
Sampling Method: Non-Probability Sample
Enrollment: 1850 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
postoperative surgical wound infection | within first week after the end of coronary artery bypass graft surgery
  postoperative surgical wound infection within first week after the end of coronary artery bypass graft surgery, classified as a superfical or deep sternal wound infection

SECONDARY OUTCOMES:
preoperative total leukocyte count | 1 day before surgery
  preoperative total leukocyte count
preoperative neutrophil count | 1 day before surgery
  preoperative neutrophil count
preoperative lymphocyte count | 1 day before surgery
  preoperative lymphocyte count
postoperative total leukocyte count | 2 hour after the end of surgery
  postoprative total leukocyte count
postoperative neutrophil count | 2 hour after the end of surgery
  postoperative neutrophil count
postoperative lymphocyte count | 2 hour after the end of surgery
  postoperative lymphocyte count
preoperative NNIS risk index | 1 day before surgery
  preoperative NNIS risk index
preoperative EuroScore | 1 day before surgery
  preoperative EuroScore
Preoperative STS | 1 day before surgery
  Preoperative STS (Society of Thoracic Surgeons risk score)
the incidence of surgical reopen with surgical wound infection | within 1 month after surgery
  the incidence of surgical reopen with surgical wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Sangmin M. Lee, MD, PhD, Principal Investigator — Samsung Medical Center; Won Ho Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea